CLINICAL TRIAL: NCT05649735
Title: EFFECTIVENESS AND SAFETY OF THE MEDICAL DEVICES LOGUSGYN ,CANDIDEP (OVULI: LOGUSGYN OVULI - FLI.000003 /CANDIDEP OVULI - FEI.000404 AND LAVENDER: LOGUSGYN Lavender - FLI.000002 / CANDIDEP LAVENDER FEI.000409) IN THE TREATMENT OF NON-SPECIFIC VULVOVAGINITIS: RANDOMISED STUDY WITH 4-ARM SEQUENTIAL DESIGN'
Brief Title: EFFICACY AND SAFETY OF OVA AND LAVAGE MEDICAL DEVICES IN THE TREATMENT OF NON-SPECIFIC VULVOVAGINITIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale del Mare (Other)
Collaborators: Erbozeta S.p.A (Unknown)
Responsible Party: Principal Investigator, Francesco Forleo, Chief, Unita Complessa di Ostetricia e Ginecologia
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ERBOLOGUS-CL-001-01
Record Dates: First submitted 2022-11-16; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-11

CONDITIONS: Vaginosis, Bacterial
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Vaginal Douching

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GROUP A- LOGUSGYN/CANDIDEP vaginal ovules, (Experimental): At baseline, eligible and PAP test negative patients were randomly assigned to receive LOGUSGYN/CANDIDEP vaginal ovules treatment for 10 consecutive days.
  Interventions: Device: Logusgyn ovules
- GROUP B- LOGUSGYN/CANDIDEP lavander (Experimental): At baseline, eligible and PAP test negative patients were randomly assigned to receive LOGUSGYN/CANDIDEP lavender treatment for 10 consecutive days.
  Interventions: Device: Logusgyn Lavander
- GROUP C- vaginal irrigation with sterile saline AELAV PURLING (Placebo Comparator): At the baseline visit, eligible and PAP test negative patients were randomly assigned to receive the vaginal irrigation with sterile saline AELAV PURLING treatment for 10 consecutive days.
  Interventions: Other: Placebo
- GROUP D- Patients pap test positive (Experimental): Patients eligible at baseline and PAP test positive will be assigned to GROUP D and treated for 10 days with sterile saline-based vaginal irrigation (Placebo/control group) AELAV PURLING- Subsequently after the initial 10-day treatment they will be randomised into two further groups, E and F, and treated for 30 days with: GROUP E- LOGUSGYN/CANDIDEP vaginal ova, GROUP F- LOGUSGYN/CANDIDEP vaginal ova, + LOGUSGYN/CANDIDEP lavage, and treated for 30 days with: GROUP E- LOGUSGYN/CANDIDEP vaginal ova, GROUP F- LOGUSGYN/CANDIDEP vaginal ova, + LOGUSGYN/CANDIDEP douche
  Interventions: Device: Logusgyn ovules; Device: Logusgyn Lavander

INTERVENTIONS:
Device: Logusgyn ovules — LOGUSGYN ovules is a CE certified Class I medical device, according to MD Directive 93/42 / EEC as amended by Directive 2007/47 / EC, manufactured by ERBOZETA S.p.a. designed for its intended use. It consists of a vaginal ova dressing for topical use containing tindalised cultures, Guar fibre, Lactic acid and Calendula.
  It is supplied in a container with 10 vaginal ova. For this study, LOGUSGYN/CANDIDEP ova/wash will be packaged according to good manufacturing practice and local regulatory requirements and will be labelled in accordance with local regulatory requirements and according to GMP Annex 13.
  Arms: GROUP A- LOGUSGYN/CANDIDEP vaginal ovules,; GROUP D- Patients pap test positive
Device: Logusgyn Lavander — LOGUSGYN lavage is a CE certified class I medical device, according to MD Directive 93/42 / EEC as amended by Directive 2007/47 / EC, manufactured by ERBOZETA S.p.a. designed for its intended use. It consists of a gynaecological lavage dressing containing Chlorhexidine 0.2% and tindalised ferments, lactic acid, bisabolol.
  It is supplied in a container with 5 vaginal douches.
  For this study, LOGUSGYN/CANDIDEP ova/wash will be packaged according to good manufacturing practice and local regulatory requirements and will be labelled in accordance with local regulatory requirements and according to GMP Annex 13.
  Arms: GROUP B- LOGUSGYN/CANDIDEP lavander; GROUP D- Patients pap test positive
Other: Placebo — Sterile saline solution
  Other Names: Vaginal irrigation with sterile saline AELAV PURLING
  Arms: GROUP C- vaginal irrigation with sterile saline AELAV PURLING

SUMMARY:
To evaluate and compare the efficacy, activity and tolerability of a vaginal ova formulation containing tindalised cultures (Lactobacillus casei, Lactobacillus acidophilus, Lactobacillus plantarum, Streptococcus thermophilus) (LOGUSGYN/CANDIDEP OVULES) and in vaginal lavage (LOGUSGYN/CANDIDEP LAVENDER) in patients with nonspecific vulvovaginitis compared to sterile saline-based vaginal irrigation (AELAV PURLING). The primary efficacy endpoint is based on the percentage of patients with therapeutic success, defined as resolution of signs and symptoms of vaginitis (total symptom score <4) at the end of treatment. For the overall assessment of clinical outcomes (resolution, improvement or failure): outcomes at the end of treatment will be considered. The treatment outcome will be measured after 5 days (V2) and after 10 days of treatment (V3) for groups A, B and C Also for group D (later, with a second randomisation, divided into groups E and F) the primary endpoint will be the same as for groups A, B, C at the visit after 30 days of treatment (V4) The treatment outcome will be measured after 5 days (V2) (after 10 days (V3) of treatment the SPT result will be re-evaluated and will be included in the secondary endpoints). The evolution of signs and symptoms of vaginitis is defined as the percentage of patients with resolution (overall score 4), improvement (decrease in overall score from baseline of 50%) or failure (decrease in overall score <50%).

Ninety-one adult female subjects (aged 18-65 years) with a diagnosis of vulvovaginitis and the presence of at least two subjective symptoms and two objective signs (at least moderate) of vaginal inflammation were recruited.

The study was planned with a randomised, controlled, parallel-group sequential design to test a vaginal ova formulation containing tindalised cultures (Lactobacillus casei, Lactobacillus acidophilus, Lactobacillus plantarum, Streptococcus thermophilus) (LOGUSGYN/CANDIDEP OVULES) and vaginal douches (LOGUSGYN/CANDIDEP LAVENDER) in patients with non-specific vulvovaginitis to control treatment (AELAV PURLING- vaginal irrigation with sterile saline). The sequential design involves a first phase with randomisation into 4 groups (A, B, C, D) followed by a second randomisation of group D (patients with vulvovaginitis and positive for HPV at PAP test) into two subgroups (E and F). The primary efficacy endpoint is based on the resolution of vulvovaginitis signs and symptoms (total SPT symptom score at the end of the first Phase I treatment period (after 5 days of treatment) for groups A, B, C and D). For the overall assessment of clinical outcomes (resolution, improvement or failure): results at the end of treatment after 10 days (V3) will be considered as secondary endpoints. Phase II will always have the resolution of vulvovaginitis signs and symptoms (total SPT symptom score f4 at the end of treatment at 30 days (V4)) as the primary endpoint, compared to Phase I results in group D.

The protocol involves 4 visits per patient over 10 days for the groups.

For groups E and F only the visit at V4 after 30 days of treatment. At visit 1 (0 days, baseline visit), patients will have to sign a written informed consent before performing any procedure. Subjects will be screened for study eligibility, verifying that all inclusion criteria and no exclusion criteria are met. At V1, the investigator will collect demographic and anamnestic data and perform a vaginal swab; in case of specific growth of pathogenic organisms, patients will be treated after the 5-day follow-up visit with antibiotics or antimycotics according to the result of the antibiogram. Delivery of the information note to the GP and the study and treatment information sheet to the patient. The investigator will then assess subjective symptomatology (burning, pain, itching, vaginal dryness, dyspareunia and dysuria) Objective symptomatology (leucorrhoea, vulvar erythema, vulvar oedema and presence of abrasion/erosion) Vaginal PH PAP test. Patients will report their degree of satisfaction with the treatment using a 5-point semiquantitative scale. Patients will be interviewed to monitor adherence to the study protocol and symptom trends during the 10-day study period (groups A, B, C and D) and at 30 days (groups E, F) The safety and tolerability of the treatments will be assessed by reporting any local and anticipated adverse events

ELIGIBILITY:
Inclusion criteria:

* Signed written informed consent
* Subjects diagnosed with vulvovaginitis
* Presence of at least two subjective symptoms and two objective signs (at least moderate) of vaginal inflammation. Vaginal inflammation will be assessed on six subjective symptoms (burning, pain, itching, vaginal dryness, dyspareunia and dysuria and four objective signs (leucorrhoea, vulvar erythema, vulvar oedema and presence of abrasion/erosion)
* The patient is able to read and understand the language and content of the study material, understand the requirements for follow-up visits, willing and able to provide information at scheduled assessments and willing and able to fulfil the requirements of the study
* PAP positive patients were allocated to group D

Exclusion Criteria:

* Persons who do not meet the inclusion criteria
* Patients who do not sign the informed consent form
* Other gynaecological diseases (in addition to cervicovaginitis), immunosuppressive diseases (i.e. HIV infection) or who are immunocompromised for reasons such as corticosteroid therapy, chemotherapy, anti-angiogenic agents or immunosuppressants
* Patients being treated with antibiotics, anti-inflammatory agents, analgesics, antineoplastic or immunosuppressive drugs within 10 days prior to inclusion in the study
* History of connective tissue disease, e.g. systemic lupus erythematosus, systemic sclerosis, Sjogren's syndrome or mixed connective tissue disease
* Known allergy to any component of the device
* Subjects who are unable to understand informed consent or who have a high probability of noncompliance with study procedures and/or noncompletion of the study in the judgment of the investigator
* Time between last day of last menstruation and baseline visit> 16 days or ≤5 days

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 91 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-08-13 (Actual)

PRIMARY OUTCOMES:
Therapeutic success | After 5 days (V2)
  resolution of signs and symptoms of vaginitis (total symptom score <4) at the end of treatment
Therapeutic success | After 10 days of treatment (V3) for groups A, B, C and D.
  resolution of signs and symptoms of vaginitis (total symptom score <4) at the end of treatment
The evolution of signs and symptoms of vaginitis | After 5 days (V2)
  the percentage of patients with resolution (overall score ≤ 4), improvement (decrease in overall score from baseline ≥ 50%), or failure (decrease in overall score <50%)
The evolution of signs and symptoms of vaginitis | After 10 days of treatment (V3) for groups A, B, C and D.
  the percentage of patients with resolution (overall score ≤ 4), improvement (decrease in overall score from baseline ≥ 50%), or failure (decrease in overall score <50%)

SECONDARY OUTCOMES:
the change from the semi-quantitative baseline score, expressed both for individual signs and symptoms and for their sum (total symptom score, TSS) | After 5 days (V2)
the change from the semi-quantitative baseline score, expressed both for individual signs and symptoms and for their sum (total symptom score, TSS) | After 10 days of treatment (V3) for groups A, B, C and D.
Vaginal pH | After 10 days of treatment (V3) for groups A, B, C and D.
Evaluation of the pap test | After 5 days (V2)
  hpv molecular swab
Evaluation of the pap test | After 10 days of treatment (V3) for groups A, B, C and D.
  hpv molecular swab

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Forleo, yes, Principal Investigator — Erbozeta
Locations (1):
- Ospedale San Giovanni Moscati, Aversa, Campania, Italy